CLINICAL TRIAL: NCT03420651
Title: Peak Expiratory Flow Rate (PEFR) for Emergency Department Management of Acute Asthma
Brief Title: Peak Expiratory Flow Rate for Emergency Department Management of Acute Asthma Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Brian Driver, Director of Clinical Research, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-4459
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Peak Expiratory Flow Rate

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: When patients are randomized to the non-peak flow guided therapy, physicians are blinded to the peak flow values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEFR Guided Management (Experimental): Peak Expiratory Flow Rate (PEFR) Patients in this group will perform PEFR testing every 30 minutes and this data along with the National Asthma Prevention and Education Program guidelines will be considered by primary ED medical providers in the management of this group.
  Interventions: Other: Peak Expiratory Flow Rate (PEFR)
- Non-PEFR Guided Management (Experimental): Standard Clinical Judgement Patients in this group will receive management based on primary medical provider's clinical judgement.
  Interventions: Other: Standard Clinical Judgement

INTERVENTIONS:
Other: Peak Expiratory Flow Rate (PEFR) — PEFR values and the National Asthma Prevention and Education Program guidelines will be used by providers in the management of these patients.
  Arms: PEFR Guided Management
Other: Standard Clinical Judgement — Providers will use physical exam and standard clinical judgement to guide management.
  Arms: Non-PEFR Guided Management

SUMMARY:
Patients presenting to the emergency department with acute asthma exacerbation will be assigned to peak-expiratory flow rate (PEFR) guided management and non-PEFR guided management.

DETAILED DESCRIPTION:
It is common practice to use peak-expiratory flow rate (PEFR) as an indicator of severity in patients that present with acute asthma exacerbation. There is, however, little data supporting this practice.

A recent Canadian 20 site prospective observational cohort study of 805 ED patients with acute asthma exacerbation concluded PEFR was not useful in predicting need for hospitalization or relapse following discharge.

As this was a cohort observational study, the conclusions that can be drawn are limited by the lack of randomization and control; it is necessary to conduct a randomized controlled trial to quantify how much time is expended caring for these patients, and gather safety data.

This is important because no studies have quantified differences in resource utilization based on PEFR-guided management compared to non-PEFR-guided management. It is possible physicians following PEFR-guided management use comparatively more resources, such as nebulizer treatments and hospitalization, in order to treat low PEFR values in patients they would have otherwise discharged based on clinical judgement alone. If outcomes are not affected by non-PEFR-guided management, it may reduce resource utilization to avoid using PEFR-guided management.

The investigators seek to determine if PEFR-based management and non-PEFR-based management perform similarly in guiding ED management of acute asthma exacerbations. Specifically, they seek to determine if the proportion of patients with no or mild asthma symptoms at 150 minutes after enrollment arrival is similar in the two groups.

At 150 minutes, it is expected that approximately 80% of patients will have no or mild asthma symptoms in both groups. When comparing the proportion of patients between the two groups, a confidence interval less than 20% wide (10% on either side of the point estimate) is desired. Therefore, goal enrollment is 110 patients per group.

This study will only include patients who are discharged from the ED. Patients who are enrolled and then eventually admitted to the hospital will be tabulated but excluded from the analysis.

Statistical analysis will compare the difference in the proportion of patients who achieve the primary outcome between groups, with the associated 95% confidence interval. Secondary outcomes will be presented descriptively; depending on the final distribution of the data, the investigators will present the means or medians of the data with the associated difference in mean/median with the associated 95% confidence intervals

ELIGIBILITY:
Inclusion Criteria:

* Presumed diagnosis of asthma, requiring at least 2 nebulized albuterol treatments
* Presenting with acute asthma exacerbation defined as acute or subacute episodes of progressively worsening shortness of breath, cough, wheezing, and chest tightness, or some combination of these symptoms
* Start of enrollment process must occur within 15 minutes of being roomed in the ED
* Working phone number and willingness to be contacted at least 72 hours following encounter

Exclusion Criteria:

* Prisoner or in custody
* Pregnant
* Known diagnosis of COPD
* Co-morbid medical conditions that patient is seeking treatment for concurrently
* Non-English speaking
* Unable to provide informed consent
* In the resuscitation bay or on non-invasive positive pressure ventilation (NPPV)

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Adequate control of asthma symptoms within 150 minutes | 150 minutes
  Proportion of patients reporting no or mild asthma symptoms at 150 minutes after enrollment

SECONDARY OUTCOMES:
Hospitalization during index encounter | 12 hours
  Rate of hospitalization in both groups directly from initial ED encounter
ED Length of Stay | 12 hours
  Time elapsed from when the patient is roomed until the time the MD places discharge order, by review of the Electronic Medical record by a blinded abstractor.
Number of nebulized treatments with short-acting beta antagonists (SABA) | 12 hours
  This is defined as the number of nebulized treatments received in the emergency department during the encounter, by review of the Electronic Medical record by a blinded abstractor.
Relapse following discharge within 72 hours | 72 hours
  Each patient will be assessed via chart review and telephone follow up to see if they visited an ED or urgent care for asthma symptoms during the 72 hour time frame. Rates of relapse will be compared between the two treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No